CLINICAL TRIAL: NCT02823808
Title: Effect of Alogliptin/Pioglitazone on the Preservation of Long-term Beta-cell Function After Early Intensive Diabetes Treatment
Brief Title: Effect of Alogliptin/Pioglitazone on the Preservation of Long-term Beta-cell Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Takeda (Industry); Kyung Hee University Hospital at Gangdong (Other); Bucheon St. Mary's Hospital (Other); Korea University Guro Hospital (Other); Ajou University School of Medicine (Other); Inha University Hospital (Other); Kangbuk Samsung Hospital (Other); Seoul Medical Center (Other)
Responsible Party: Principal Investigator, Jeong-taek Woo, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KNDP_IIT_2016_01
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALO+PIO (Experimental): Group who takes Alogliptin 25mg+Pioglitazone 15mg, once daily.
  Interventions: Drug: NESINA ACT TAB. 25/15mg
- GMPD+MET (Active Comparator): Group who takes Glimepiride 2mg+Metformin 500mg, once daily.
  Interventions: Drug: AMARYL-M TAB. 2/500mg

INTERVENTIONS:
Drug: NESINA ACT TAB. 25/15mg — Alogliptin/Pioglitazone 25/15mg will be administered to the group once a day in a fixed dose on a fixed schedule for 104 week.
  Arms: ALO+PIO
Drug: AMARYL-M TAB. 2/500mg — Glymepiride/Metformin 2/500mg will be administered to the group once a day in a fixed dose on a fixed schedule for 104 week.
  Arms: GMPD+MET

SUMMARY:
All subjects will be randomized as Alo/Pio combo group (intervention) or Glim/Met combo group (control) after intensive COAD treatment based on identical protocol.

* All subject will be managed with once daily, fixed dose, single tablet treatment based on the study protocol, and followed-up for 104 weeks.
* Any group of subjects who fail to reach glycemic target with single tablet treatment, subject will be treated with rescue medication and stopped regular observation.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus patients
* Patient who had been diagnosed within the previous 12 months with HbA1c levels of 8.0-12.0%, did not have a medical history related to diabetes, and did not display proliferative retinopathy

Exclusion Criteria:

* The use of weight-lowering drugs, any investigational blood-glucose or lipid-lowering agent (other than statins or ezetimibe) within the past 3 months
* Previous treatment with systemic corticosteroids or a change in dosage of thyroid hormones in the previous 6 weeks
* The use of insulin within the 3 months prior to screening
* Others

Ages: 26 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative treatment failure (HbA1c≥7.0%) rate for glycemic control | 104 weeks from randomization

SECONDARY OUTCOMES:
Change in HbA1c | 104 weeks from randomization
Change in Fasting Blood Sugar | 104 weeks from randomization
Change in Glycoalbumin | 104 weeks from randomization
Change in insulin sensitivity (HOMA2%S) | 104 weeks from randomization
Change in insulin sensitivity (HOMA2%B) | 104 weeks from randomization
Change in proinsulin | 104 weeks from randomization
Change in glucagon | 104 weeks from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-taek Woo, Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyunghee University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No